CLINICAL TRIAL: NCT05903937
Title: Hepatic Arterial Infusion of Autologous Tumor Infiltrating Lymphocytes Preconditioned With Percutaneous Hepatic Perfusion With Melphalan in Patients With Melanoma and Liver Metastases
Brief Title: Locoregional Administration of TIL and Lymphodepletion in Patients With Melanoma and Liver Metastases
Acronym: HAITILS-PHP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-006126-32
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Uveal Melanoma; Metastatic Cutaneous Melanoma
Keywords: TIL; ACT; PHP
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Melphalan; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous tumor infiltrating lymphocytes (TIL) (Experimental)
  Interventions: Drug: Autologous Tumor Infiltrating Lymphocytes; Drug: Melphalan; Drug: Interleukin-2

INTERVENTIONS:
Drug: Autologous Tumor Infiltrating Lymphocytes — Administered via hepatic arterial infusion (HAI)
Drug: Melphalan — Administered via isolated hepatic perfusion
Drug: Interleukin-2 — low-dose, administered s.c.

SUMMARY:
Evaluate the safety and tolerability of treatment with autologous tumor infiltrating lymphocytes (TIL) administered via hepatic arterial infusion and preconditioning with percutaneous hepatic perfusion in patients with liver metastases (but not restricted to) of malignant melanoma

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide written informed consent and comply with study procedures. Written informed consent must be signed and dated before the start of specific protocol procedures.
* Patient must have a histologically/cytologically confirmed diagnosis of:
* stage IV uveal melanoma with or without any previous systemic therapy OR
* stage IV cutaneous melanoma with confirmed progression following at least one or two prior systemic therapies including a programmed cell death protein-1 (PD-1) inhibitor with or without a CTLA-4 inhibitor; and if BRAF V600 mutation-positive, also a BRAF inhibitor or a BRAF inhibitor in combination with a MEK inhibitor.
* Measurable disease by computed tomography (CT) per RECIST 1.1 criteria with at least one target lesion identified in the liver and where the distribution pattern of metastasis is predominantly engaging the liver as judged by the investigator.
* At least one resectable lesion in the liver (or aggregate of lesions resected) of a minimum size of 0.5 cm in diameter post- resection to generate TILs.
* ECOG performance status of 0 - 1.

Exclusion Criteria:

* Life expectancy of less than 3 months.
* Reduced renal function defined as S-Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockroft and Gault formula.
* Reduced hepatic function (defined as ASAT, ALAT, bilirubin > 3*ULN and PK- INR > 1.5) or medical history of liver cirrhosis or portal hypertension.
* Hemoglobin <90 g/L or platelets <100x109/L or neutrophils <1.5x109/L
* Use of live vaccines four weeks before or after the start of study.
* Infection of human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C.
* Active autoimmune disease.
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Concomitant therapy with any other anti- cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs.
* Has a known additional malignancy of other diagnosis that is progressing or requires active treatment.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 5 years
  Graded according to Common Terminology Criteria for Adverse Events version 5.0

SECONDARY OUTCOMES:
Objective response rate | 5 years
  Defined as the proportion of patients with a best overall response of partial response or better defined by RECIST 1.1
Progression-free survival | 5 years
  Defined as the time from inclusion to objective tumor progression (determined by RECIST 1.1), or death due to any cause, whichever occurred first.
hepatic Progression-free survival | 5 years
  Defined as the time from inclusion to objective tumor progression in the liver (determined by RECIST 1.1), or death due to any cause, whichever occurred first.
Duration of response | 5 years
  Defined as the time from the first documented response and the date of the first documented tumor progression, death, or the last tumor assessment that occurred before subsequent therapy.
Overall survival | 5 years
  Defined as the time from inclusion to the date of death due to any cause
Evaluation of Tolerability | 5 years
  Defined as the proportion of patients included that receive PHP and TIL

IPD SHARING:
Plan to Share IPD: No